CLINICAL TRIAL: NCT01818544
Title: A Phase IIa, Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Safety and Efficacy of 28 Day Oral Administration of BAY85-8501 in Patients With Non-Cystic Fibrosis Bronchiectasis
Brief Title: Safety and Efficacy of Oral BAY85-8501 in Patients With Non-CF (Cystic Fibrosis) Bronchiectasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16359; 2012-004491-18 (EudraCT Number)
Record Dates: First submitted 2013-03-08; First posted 2013-03-26 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Bronchiectasis
Keywords: Elastase Inhibition
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BAY85-8501 (Experimental)
  Interventions: Drug: BAY85-8501
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY85-8501 — BAY85-8501 (1.0 mg, 2 tablets each 0.5 mg) will be administered orally once daily in the morning
  Arms: BAY85-8501
Drug: Placebo — Placebo (1.0 mg, 2 tablets each 0.5 mg) will be administered orally once daily in the morning
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of 28 day oral administration of BAY85-8501 versus placebo in subjects with non-CF Bronchiectasis (BE).

The secondary objectives are to examine the effect of BAY85-8501 on pulmonary function, biomarkers of inflammation and tissue damage, and the impact on overall health and perceived well-being and to evaluate the pharmacokinetics of BAY85-8501.

ELIGIBILITY:
Inclusion Criteria:

* Proven and documented diagnosis of non-CF (cystic fibrosis) idiopathic or post-infectious BE (bronchiectasis) by computed tomography (CT) scan [conventional high resolution CT is considered the standard], including 2 or more lobes and dilated airways compatible with BE at initial diagnosis
* Stable pulmonary status as indicated by the forced, expired volume in 1 second (FEV1) percent predicted ≥30% and <90% (post-bronchodilator)
* Stable (i.e., no dose change) regimen of standard BE treatment administered at least for 4 weeks prior to screening
* Cough on most days

Exclusion Criteria:

* Forced, expired volume in 1 second <30% or ≥90% predicted (post-bronchodilator)
* Recent significant hemoptysis (≥300 mL or requiring blood transfusion) in the preceding 4 weeks before screening (and during the screening period)
* Known cystic fibrosis and/or documented chronic bronchial asthma
* Active allergic bronchopulmonary aspergillosis (ABPA)
* Diagnosis of common variable immunodeficiency (CVID)
* Systemic or inhaled antibiotic treatment within 4 weeks prior to screening
* Treatment of an exacerbation within 4 weeks prior to screening
* Systemic corticosteroids at >10 mg/day prednisolone equivalent for >2 weeks within 4 weeks prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2013-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number Of Subjects Who Need To Discontinue Study Medication Due To Findings In Physical Examination | From start of study treatment up to follow up visit (28 days after last dose)
Change From Baseline in Systolic Blood Pressure At Days 7, 14, 21, 28, 56 | Baseline (Day 1), Day 7, 14, 21, 28, 56
Change From Baseline in Diastolic Blood Pressure At Days 7, 14, 21, 28, 56 | Baseline (Day 1), Day 7, 14, 21, 28, 56
Change From Baseline in Heart Rate At Days 7, 14, 21, 28, 56 | Baseline (Day 1), Day 7, 14, 21, 28, 56
Number of Subjects With new Abnormal (Pathologic) Electrocardiogram (ECG) Findings From Baseline to Day 28 | Baseline (Day 1), Day 7, 14, 21, 28
Number of Subjects who Show Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Total Bilirubin (TB) Abnormalities in Their Safety Lab Assessment | Baseline (Day 1), Day 7, 14, 21, 28, 56
Number of Subjects With Drug Related Adverse Events as a Measure of Safety And Tolerability | Baseline (Day 1), Day 7, 14, 21, 28, 56

SECONDARY OUTCOMES:
Change From Baseline in Pulmonary Function Test Forced Expired Volume in 1 Second (FEV1) At Days 7, 14, 21, 28, 56 | Baseline (Day 1), Day 7, 14, 21, 28, 56
Change From Baseline in Pulmonary Function Test Forced Vital Capacity (FVC) at Days 7, 14, 21, 28, 56 | Baseline (Day 1), Day 7, 14, 21, 28, 56
Change From Baseline in Pulmonary Function Test Forced Expiratory Flow Over the Middle Half of Subject's Forced Vital Capacity (FVC) (FEF2575) at Days 7, 14, 21, 28, 56 | Baseline (Day 1), Day 7, 14, 21, 28, 56
Change From Baseline in Total Score on St. George's Respiratory Questionnaire (SGRQ) at Day 28 and 56 | Baseline (Day 1), Day 28 and 56
Change From Baseline in 24 Hours Sputum Weight at Day 28 | Baseline (Day 1), Day 28
Change From Baseline of Biomarkers in Sputum at Days 14, 28, 56: Alpha1 Antitrypsin Human Neutrophil Elastase (A1AHNE) Complex, Interleukin-8(IL-8) | Baseline (Day 1), Day 14, 28 and 56
Change From Baseline of Biomarkers in Sputum at Days 14, 28, 56: Neutrophil cell Count | Baseline (Day 1), Day 14, 28 and 56
Change From Baseline of Human Neutrophil Elastase (NE) Activity in Sputum at Days 14, 28, 56 | Baseline (Day 1), Day 14, 28 and 56
Change From Baseline of Human Neutrophil Elastase (NE) Concentration in Sputum at Days 14, 28, 56 | Baseline (Day 1), Day 14, 28 and 56
Change From Baseline of Biomarkers in Blood at Days 14, 28, 56: C-reactive Protein | Baseline (Day 1), Day 14, 28 and 56
Change From Baseline of Biomarkers in Blood at Days 14, 28, 56: Interleukin-8 (IL8) | Baseline (Day 1), Day 14, 28 and 56
Change From Baseline of Biomarkers in Blood at Days 14, 28, 56: Neutrophil cell Count | Baseline (Day 1), Day 14, 28 and 56
Change From Baseline of Biomarkers in Urine At Days 14, 28, 56: Creatinine | Baseline (Day 1), Day 14, 28 and 56
Change From Baseline of Biomarkers in Urine at Days 14, 28, 56: Desmosine | Baseline (Day 1), Day 14, 28 and 56
Change From Baseline of Biomarkers in Urine at Days 14, 28, 56: Normalized Desmosine Value to Creatinine | Baseline (Day 1), Day 14, 28 and 56

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (33):
- France (2):
  - Nice
  - Perpignan
- Germany (9):
  - Donaustauf, Bavaria
  - Rüdersdorf, Brandenburg
  - Hamburg, Hamburg
  - Hanover, Lower Saxony
  - Leipzig, Saxony
  - Großhansdorf, Schleswig-Holstein
  - Kiel, Schleswig-Holstein
  - Lübeck, Schleswig-Holstein
  - Jena, Thuringia
- Italy (6):
  - Orbassano, Torino
  - Genova
  - Milan
  - Napoli
  - Padua
  - Siena
- Spain (4):
  - Badalona, Barcelona
  - Salt, Girona
  - Madrid, Madrid
  - Majadahonda, Madrid
- United Kingdom (12):
  - Southampton, Hampshire
  - Cottingham, Humberside
  - Leicester, Leicestershire
  - Liverpool, Merseyside
  - Sheffield, South Yorkshire
  - Dundee, Tayside
  - Newcastle upon Tyne, Tyne and Wear
  - South Shields, Tyne and Wear
  - Wolverhampton, West Midlands
  - Bradford, West Yorkshire
  - Glasgow
  - London

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/